CLINICAL TRIAL: NCT02049203
Title: A Phase Ib Randomized, Placebo-controlled, Double-blinded Study Evaluating the Safety of Ataciguat (HMR1766) in Patients With Moderate Calcific Aortic Valve Stenosis
Brief Title: Safety of Ataciguat in Patients With Moderate Calcific Aortic Valve Stenosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jordan D. Miller, Ph.D. (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Sanofi-Synthelabo (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Jordan D. Miller, Ph.D., Assistant Professor of Surgery, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-005387; UL1RR024150 (NIH)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — 5-chloro-2-(5-chlorothiophene-2-sulfonylamino)-N-(4-(morpholine-4-sulfonyl)phenyl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo gel capsule, dosage matches number of Ataciguat capsules for each respective dose, capsules taken once daily with breakfast for 14 consecutive days.
  Interventions: Drug: Placebo
- Ataciguat (Active Comparator): Ataciguat, orally administered gel capsule, 50, 100, or 200 mg, once per day with breakfast for 14 consecutive days
  Interventions: Drug: Ataciguat

INTERVENTIONS:
Drug: Ataciguat
  Other Names: HMR1766
  Arms: Ataciguat
Drug: Placebo
  Other Names: Placebo gel capsule of identical composition to Active group, but does not have active compound.
  Arms: Placebo

SUMMARY:
This study will determine whether Ataciguat (HMR1766) is well-tolerated in patients with mild to moderate calcific aortic valve stenosis. The primary focus of these studies will be on changes in blood pressure and orthostatic tolerance (i.e., ability to stand up without passing out), and determining whether treatment with Ataciguat results in significant reductions in blood pressure in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Male or female sex
* Aortic valve area greater than 1.0 cm2 but less than 2.0 cm2
* Aortic valve calcium levels greater than 300 arbitrary units from chest CT
* Ejection fraction >50%

Exclusion Criteria:

* History of orthostatic intolerance or symptomatic hypotension
* Positive pregnancy test during screening visit
* Nitrate use or α-antagonist medication use within 24 hours
* Systolic blood pressure <110 mm Hg
* Mean systemic arterial pressure <75 mm Hg
* Severe mitral or aortic regurgitation
* Retinal or optic nerve problems
* Recent (≤30 days) acute coronary syndrome
* Oxygen saturation <90% on room air
* Congenital valve disease
* Hepatic dysfunction/elevated liver enzymes
* Prescription of drugs known to alter nitric oxide-soluble guanylate cyclase-cyclic guanosine monophosphate signaling (sildenafil, nitrates, etc.)
* History of orthostatic intolerance
* Concomitant participation in other trials at Mayo Clinic or elsewhere.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing orthostatic hypotension | Baseline - 14 days
  The primary objective of the current study is to determine whether Ataciguat (HMR1766) is well-tolerated by patients with moderate calcific aortic valve stenosis. In this particular patient population, incidence of orthostatic intolerance/symptomatic hypotension is a potential concern.
The change in blood pressure following the transition from sitting to standing | Baseline - 14 days
  The primary objective of the current study is to determine whether Ataciguat (HMR1766) is well-tolerated by patients with moderate calcific aortic valve stenosis. In this particular patient population, incidence of orthostatic intolerance/symptomatic hypotension is a potential concern. Transitioning from sitting to standing is a functional test that will allow us to examine the effects of Ataciguat on blood pressure regulation in response to a relevant orthostatic stress.
The change in blood pressure following progressive head-up tilt | Baseline - 14 days
  The primary objective of the current study is to determine whether Ataciguat (HMR1766) is well-tolerated by patients with moderate calcific aortic valve stenosis. In this particular patient population, incidence of orthostatic intolerance/symptomatic hypotension is a potential concern. Tilt table testing will allow us to examine the effects of Ataciguat on blood pressure regulation in response to a tightly controlled orthostatic stress.
Subject self-reports of light-headedness/orthostatic intolerance during the standing test and the head-up tilt testing | Baseline - 14 days
  The primary objective of the current study is to determine whether Ataciguat (HMR1766) is well-tolerated by patients with moderate calcific aortic valve stenosis. In this particular patient population, incidence of orthostatic intolerance/symptomatic hypotension is a potential concern. Evaluating subject perceptions of light-headedness/orthostatic intolerance will help us to understand the relationship between changes in blood pressure and changes in symptoms in this patient population before and after treatment with Ataciguat.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Miller, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Zhang B, Enriquez-Sarano M, Schaff HV, Michelena HI, Roos CM, Hagler MA, Zhang H, Casaclang-Verzosa G, Huang R, Bartoo A, Ranadive S, Joyner MJ, Pislaru S, Nkomo VT, Kremers WK, Araoz PA, Singh G, Walters MA, Hawkinson J, Cunningham KY, Sung J, Dunagan B, Ye Z, Miller JD. Reactivation of Oxidized Soluble Guanylate Cyclase as a Novel Treatment Strategy to Slow Progression of Calcific Aortic Valve Stenosis: Preclinical and Randomized Clinical Trials to Assess Safety and Efficacy. Circulation. 2025 Apr;151(13):913-930. doi: 10.1161/CIRCULATIONAHA.123.066523. Epub 2025 Feb 24. PMID 39989354